CLINICAL TRIAL: NCT04389788
Title: Efficacy and Safety of Combined Microneedling With Topical Glutathione Versus Carboxy Therapy in Treatment of Patients With Periorbital Hyperpigmentation
Brief Title: Treatment of Patients With Periorbital Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Abdelhamed, Lecturer of Dermatology, Venereology & Andrology, Sohag University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Sohagu309
Record Dates: First submitted 2020-05-04; First posted 2020-05-15 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Periorbital Hypermelanosis
Keywords: Periorbital hypermelanosis; Carboxy therapy; Microneedling; Topical Glutathione

STUDY DESIGN:
Intervention Model Description: Patients with periorbital hyperpigmentation will be treated using Carboxy theraby method at right side of face followed by microneedling using dermapen will be at left side of face.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and the outcome assessors were blinded to the type of treatment which was done in each eye
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rt Eye (Active Comparator): The right eye of the patients received carboxy therapy for 6 sessions every 2 weeks. The used device is locally manufactured by a national company for esthetic and dermatological devices. Carbon dioxide gas was subcutaneously injected at the lateral one-third of each eye lid (5 cc gas in each puff according to standardized flowmetry) using insulin syringe. Compression of the injected area will be avoided to prevent rapid leakage of the gas.
  Interventions: Device: carboxy therapy
- Lt Eye (Active Comparator): The left eye of the same patients received microneedling with topical glutathione for 6 sessions every 2 weeks. Microneedling was done with Derma pen which is automatic and rechargeable device (vibrating frequency : 6500-10000 r/m , vibration speed level 5 , model :Ultima A6 , company : Dr ,pen and country : Korea). Needle length is adjustable from 0.25 mm to 0,5 mm.Needles number : 36 .Then, Patient was subjected to topical glutathione about 0.25 ml (vial : 600mg/5ml).
  Interventions: Device: Dermapen with topical glutathione

INTERVENTIONS:
Device: carboxy therapy — 6 sessions of carboxy therapy every 2 weeks
  Arms: Rt Eye
Device: Dermapen with topical glutathione — 6 sessions of Dermapen microneedling with topical glutathione every 2 weeks
  Arms: Lt Eye

SUMMARY:
Periorbital hyperpigmentation (POH) is a common condition in dermatology practice. Periorbital hyperpigmentation is defined as bilateral, round, homogeneous pigmented macules.The etiology of POH is multifactorial including genetic and enviromental factors. Many treatment options are avaiblabe with variable efficacy and safety in different patients. Therefore, the investigator's study aims to evaluate the efficacy and safety of combined microneedling with topical Glutathione versus Carboxy Therapy in treatment of patients with periorbital hyperpigmentation.

DETAILED DESCRIPTION:
Periorbital hyperpigmentation (POH) is a common skin condition which has a great negative effect on the patient quality of life. Many factors contribute in the pathogensis of POH which lead to developement of several treatment options with no treatment option has a great sucess in improving the POH and patient quality of life. Our current study tries to explore the efficacy and safety between 2 treatment methods in a split face study.

Microneedling is a process of making small punctres into the skin through small needles by device which is called a Dermapen. This microneedling method is beleived to be associated with improving the skin quality through increased collagen. This microneedling will be followed by topical application of glutathione which is a commong antioxidant with whitening effects.

Carboxy therapy is a new emerging treatment option in many dermatological diseases. It will be used in POH patients as it will be able to increase blood flow in periorbital area and improve the skin qulaity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Periorbital hyperpigmentation

Exclusion Criteria:

* Pregnancy and lactation .
* Allergy, hypersensitivity to the formulations to be used in the study.
* Any other cutaneous or systemic disease.
* Patient who had taken any other treatment (laser, dermabrasion) on the affected region performed less than 6 months prior to the beginning of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Change of periorbital hyperpigmentation through photo evaluation | Baseline, before 3rd session, before 5th session, 1 month after end of treatment, 2 months after end of treatment
  High-resolution photographs of both sides of the face were taken. Using a physician visual analog scoring system, 2 independent blinded dermatologists will rate the patient's overall aesthetic improvement as follows 1 (worse), 2 (no change), 3 (<30%), 4 (30-60%), and 5 (>60%)
Change of periorbital hyperpigmentation through dermoscopy evaluation | Baseline, before 3rd session, before 5th session, 1 month after end of treatment, 2 months after end of treatment
  Dermoscopic evaluation was done using dermalite connection kit for Samsung galaxy. 2 independent blinded dermatologists will rate the patient's overall aesthetic improvement as follows
  * Vasculature improvement (No 0, Yes 1) & percent of improvement.
  * Pigmentation improvement (No 0, Yes 1) & percent of improvement.
  * Skin improvement like atrophy and exaggerated skin markings (No 0, Yes 1) & percent of improvement.
Change of the patient satisfaction evaluation: scale | Baseline and 1 month after end of treatment
  The patients were asked to evaluate their own level of satisfaction after they completed the study on a 1-3 scale: 1 = slightly satisfied, 2 = moderately satisfied, and 3 = well satisfied
Change of periorbital hyperpigmentation into another skin problem through safety evaluation | Baseline, before 3rd session, before 5th session, 1 month after end of treatment, 2 months after end of treatment
  Safety evaluation to detect precentage of side effects reported either by the patient or by the physician.

SECONDARY OUTCOMES:
The Dermatology Life Quality Index questionnaire | Baseline, before 3rd session, before 5th session,
  The Dermatology Life Quality Index questionnaire (DLQI) is 10 questions were asked to the patients and score is 0-3 for each question. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: At the end of study july 2020.

REFERENCES:
- [Derived] Assaf HA, Ahmed D, Abdelhamed A. Efficacy and Safety of Carboxytherapy versus Combined Microneedling with Topical Glutathione in the Treatment of Patients with Periorbital Hyperpigmentation: An Evaluator-Blind, Split-Face, Controlled Pilot Clinical Trial. Indian J Dermatol. 2022 Sep-Oct;67(5):504-511. doi: 10.4103/ijd.ijd_394_21. PMID 36865870